CLINICAL TRIAL: NCT02220114
Title: Acceptability Study of a New Paediatric Form of Vigabatrin in Infants and Children With Infantile Spasms or Pharmacoresistant Partial Epilepsy. Observational, Descriptive, Open-label, Multi-centric, Non-randomized Study
Brief Title: Acceptability Study of a New Paediatric Form of Vigabatrin in Infants and Children With Infantile Spasms or Pharmacoresistant Partial Epilepsy
Acronym: SoluWest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orphelia Pharma (Industry)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Hospices Civils de Lyon (Other); National Research Agency, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TGO-VGB-III-01
Record Dates: First submitted 2014-08-14; First posted 2014-08-19 (Estimated); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Infantile Spasms
Keywords: Infantile spasms; vigabatrin; soluble tablets; acceptability; adherence; pharmacokinetics
MeSH Terms: conditions — Spasms, Infantile

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vigabatrin: Vigabatrin new ST formulation then Sabril® (Other): Sabril®: sachet for oral solution 500 mg, 50 to 100mg/Kg/day, twice a day, 14 days.
  Vigabatrin new ST formulation: Soluble tablets 100 or 500 mg, 50 to 100mg/Kg/day, twice a day, 12 weeks.
  Interventions: Drug: Vigabatrin: Vigabatrin new ST formulation then Sabril®

INTERVENTIONS:
Drug: Vigabatrin: Vigabatrin new ST formulation then Sabril® — * first "treatment" phase (V1/D1-V3/D84), in which patients already under Sabril® "granules for oral solution" and naive patients start the new ST formulation; patients already under Sabril® will start at the same dose and regimen as their usual Sabril®. Dose and regimen for naive patients will be chosen according to SPC.
  * second "treatment" phase (V3/D84-V4/D98) in which the patient is switched to Sabril® "granules for oral solution" (supplied by sponsor) for 15 days at the same dose as under the new ST formulation.
  Dose and treatment regimen should be maintained as in first treatment phase.
  - At V4/D98, patients who received Sabril® "granules for oral solution" (supplied by sponsor) continue with marketed Sabril® treatment (or switches to another AED, according to the natural evolution of the patient's condition and upon investigator decision).

SUMMARY:
The sponsor is developing a new paediatric formulation of vigabatrin to better adjust the dose to body weight and to limit waste of unused drug. The currently marketed vigabatrin (Sabril™) form only exists as 500 mg film coated tablets (for adults and children above 6 years) and 500 mg granules for oral solution sachets (for infants and children below 6 years). Sabril™ is not adapted for administration to infants when a fraction of the sachet is needed. Manual splitting of the sachet or lengthy and error-prone dilutions are often required.

This study is a descriptive, non-randomized, open label multi-centric acceptability study in infants and children affected with infantile spasms. The primary objective is to describe the adherence to the new formulation. Secondary objectives include:

* evaluation of the palatability and user-friendliness of the new treatment,
* evaluation of the pharmacokinetic parameters of the new formulation,
* PK parameters,
* evaluation of the tolerance,
* measurement of taurine plasma levels. This study will recruit up to 40 patients with infantile spasms and pharmacoresistant partial epilepsy aged 1 month to 6 years in 23 clinical sites in France.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosed infantile spasms (IS) or pharmacoresistant partial onset seizures (POS).
* Infants > 1 month and < 6 months; infants > 6 months and < 2 years; and children > 2 years and < 6 years.
* Patients under Sabril® or naive patients.
* Patients under a twice-a-day posology of Sabril® or patients for whom vigabatrin will be given twice daily.

Non inclusion Criteria:

* Use of more than 2 other antiepileptic drugs as concomitant treatment (including steroids). Ketogenic diet can be in addition to these 2 other antiepileptic drugs.
* Subjects receiving vigabatrin through a gastric tube.
* Weight < 1.750 Kgs.
* Any planned major surgery within the duration of the trial.
* Participation in any other clinical trial within 3 months prior to V1.

Ages: 1 Month to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2014-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Individual adherence to the new Soluble Tablets (ST) formulation of Vigabatrin (VGB) using Medication Event Monitoring System (MEMS) | from V1 (day 1) to V3 (day 84), continuous assessment.
  Adherence will be assessed by measurement of the dosing history of patients using an electronic Medication Event Monitoring System (MEMS).The date and time of each opening will be recorded

SECONDARY OUTCOMES:
Adherence to the new ST formulation and to Sabril® granules for oral solution, by treatment unit accountability | VGB-ST: V1 (day 1) to V3 (day 84). Sabril®:V3 (day 85) to V4 (day 98)
  Accountability of used and unused treatment units, retrieved by the patient at V3 and V4
palatability of the new ST formulation and of Sabril® "granules for oral solution". | during 7 consecutive days: from D90 to D96 under Sabril® and from D29 to D35 under the new ST formulation
  Palatability of the treatment will be evaluated using a two face visual hedonic scale filled in by the parents and/or by the child, if feasible, on a daily basis. Each "face" of the scale will be assigned a score (1 to 2), and the average score will be calculated for the group. Palatability will be considered good if the average score for the group is at least 1.5 (out of a maximum of 2; Motte et al. 2005).
Ease of use of the new ST formulation and of Sabril® "granules for oral solution". | during 7 consecutive days: from D90 to D96 under Sabril® and from D29 to D35 under the new ST formulation.
  Ease of use will be evaluated using diaries filled by the parents or care-givers during 7 consecutive days: . Time required for preparation of both new ST formulation and Sabril® administrations will be averaged and compared, together with the global use satisfaction.
Safety and tolerance | Results of electroretinogram: when available from D1 to D126; Blood assessment: at D1 & D84; Vital signs at D1, D28, D84, D98 & D126; Adverse events, serious adverse events: evaluated for the duration of study participation (at D1, D28, D84, D98 & D126)
  VGB safety profile is well known. The new ST formulation is expected to be bioequivalent to Sabril®, and since the new formulation does not contain excipients known to have a recognized action or effect at the dose used, the safety of the new formulation should be similar to that of Sabril®. Hence no other measures specific to the new ST formulation are included in the clinical acceptability study.
pharmacokinetic parameters for the new ST formulation (1 sample). Pharmacokinetic parameters for the new ST formulation (population PK) : Area under the curve (AUC), Tmax, Cmax, T½, Ka, V/F, Cl/F | PK D84: 1 sample before treatment.
  The objective is to better characterize the developmental PK of vigabatrin during childhood.
Evaluation of the taurine plasma levels in children treated by vigabatrin. Taurine plasma concentration will be measured and a relationship between vigabatrin exposition and taurine plasma levels will be sought. | 1 sample will be drawn at V3 (day 84): just before treatment when patient is fasting.

CONTACTS AND LOCATIONS:
Overall Officials: Rima NABBOUT, Principal Investigator — Hôpital Necker Enfants Malades - APHP
Locations (12):
- France (12):
  - Service de neurologie pédiatrique - CHU, Amiens
  - Service de neurologie pédiatrique - CHU, Angers
  - Service de neuropédiatrie - CHU Pellegrin Enfants, Bordeaux
  - Service de neurologie infantile - Hôpital Salengro, Lille
  - Service de nuerologie pédiatrique - Hôpital Femme Mère Enfant, Lyon
  - Service de neurologie pédiatrique - Hôpital de la Timone, Marseille
  - Service de neurologie pédiatrique - Hôpital Necker Enfants Malades, Paris
  - Service de neuropédiatrie - Hôpital Robert Debré, Paris
  - Service de neurologie pédiatrique - Hôpital Sud, Rennes
  - Centre référent des épilepsies rares pédiatrique associé - Hôpital de Hautepierre, Strasbourg
  - Service de neuropédiatrie - Hôpital Purpan, Toulouse
  - Service de neuropédiatrie - Hôpital de Clocheville, Tours